CLINICAL TRIAL: NCT01055587
Title: Impact of Biomarkers for Early Diagnostic of Infections Following Major Abdominal Surgery and Severe Burn Injuries
Brief Title: Diagnostic of Infections Following Major Abdominal Surgery and Burn Injury
Acronym: Earlygnost
Status: Completed | Type: Observational
Sponsor: Klinikum St. Georg gGmbH (Other)
Collaborators: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Armin Sablotzki, MD, Prof. Dr. med., Klinikum St. Georg gGmbH
Other Study IDs: EK-BR-29/09-1; Stu09/0031
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Third Degree Burn; Second Degree Burn
Keywords: major abdominal surgery; severe burn injury; infection; diagnostic
MeSH Terms: conditions — Burns; Infections; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- major abdominal surgery: The investigators compare the levels of biomarkers in patients with and without complications in the early postoperative course following major abdominal surgery
- severe burn injury: The investigators compare levels of biomarkers within the first 20 days in patients with and without complications following severe burn injury

SUMMARY:
This study was designed to investigate, if new biomarkers may improve the early diagnostic of infections following major abdominal surgery and severe burn injuries.

ELIGIBILITY:
Inclusion Criteria:

* patients with major abdominal surgery (e.g. gastrectomy, hemi-/colectomy, resection of sigma or rectum, resection of liver, esophagectomy)
* patients following severe burn injury (burn surface area >= 15%)
* age >= 18 years
* informed consent

Exclusion Criteria:

* no informed consent
* emergency surgery
* immunocompromising diseases (e.g. HIV+, AIDS, Lymphoma or NonHodgkin-Lymphoma, Autoimmune-Diseases)
* pre-existing liver or renal failure
* chronic therapy with corticoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: patients who undergo major abdominal surgery Group 2: patients following severe burn injury
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2009-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
rate of infections | day 28 post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Armin R Sablotzki, MD, Principal Investigator — Klinikum St. Georg gGmbH
Locations (1):
- Klinikum St. Georg gGmbH, Leipzig, Saxony, Germany

REFERENCES:
- [Derived] Gille J, Schmidt J, Kremer T, Sablotzki A. Evaluation of MR-proANP and copeptin for sepsis diagnosis after burn injury. J Crit Care. 2019 Aug;52:149-155. doi: 10.1016/j.jcrc.2019.04.031. Epub 2019 Apr 30. PMID 31075618
- [Derived] Gille J, Ostermann H, Dragu A, Sablotzki A. MR-proADM: A New Biomarker for Early Diagnosis of Sepsis in Burned Patients. J Burn Care Res. 2017 Sep/Oct;38(5):290-298. doi: 10.1097/BCR.0000000000000508. PMID 28221298